CLINICAL TRIAL: NCT03716648
Title: Determination of the Optimal Mandibular Position During Oral Appliance Therapy With a Mandibular Advancement Device in Patients Diagnosed With Obstructive Sleep Apnea.
Brief Title: Titration of Oral Appliance Therapy: a Prospective, Randomized Cross-over Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, ethisch.comite@uza.be, prof. dr. Olivier Vanderveken, MD, PhD, University Hospital, Antwerp
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18/33/364
Record Dates: First submitted 2018-10-09; First posted 2018-10-23 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Randomized, crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Subjective titration (Active Comparator): After fitting the MAD, there is a 1-month period during which the patients get used to wearing the device and titrate the MAD based on improvement of subjective complaints. The actual mechanism of titration will be individually trained with each patient.
  Interventions: Device: subjective titration
- DISE-assisted titration (Experimental): Incremental protrusion of the mandible during drug-induced sleep endoscopy using the remotely controlled mandibular positioner until upper airway collapse at all collapsible levels is eliminated.
  Interventions: Diagnostic Test: DISE-assisted titration
- PSG-guided titration (Experimental): An overnight titration polysomnograph using the remotely controlled mandibular positioner with stepwise mandibular protrusion until respiratory events are reduced.
  Interventions: Diagnostic Test: PSG-guided titration

INTERVENTIONS:
Diagnostic Test: DISE-assisted titration — Titration of the mandibular position with the remotely controlled mandibular positioner during drug-induced sleep endoscopy.
  Arms: DISE-assisted titration
Diagnostic Test: PSG-guided titration — Titration of the mandibular position with the remotely controlled mandibular positioner during drug-induced sleep endoscopy.
  Arms: PSG-guided titration
Device: subjective titration — Titration of the mandibular position based on subjective improvement in symptoms like snoring and excessive daytime sleepiness.
  Arms: Subjective titration

SUMMARY:
In this prospective randomized cross-over trial, 3 different titration procedures will be compared:

1. titration of the mandibular advancement device (MAD) in the home setting based on both the physical limits of the patient's mandibular protrusion and the resolution of subjective complaints, as currently often used in routine clinical practice;
2. an overnight titration PSG using the remotely controlled mandibular positioner (RCMP) with stepwise mandibular protrusion until respiratory events are reduced and
3. incremental protrusion of the mandible during DISE using the RCMP until upper airway collapse at all collapsible levels is eliminated.

The aim of this study is to prospectively compare the target protrusion, as well as the treatment outcome in terms of treatment efficacy, of the 3 different titration protocols.

DETAILED DESCRIPTION:
After inclusion, each patient will undergo three different titration procedures of the protrusive mandibular position or target protrusion for the MAD treatment, in a randomized order: subjective titration, titration during DISE, titration during PSG.

1. Subjective titration:

   After fitting the MAD, there is a 1-month period during which the patients get used to wearing the device and titrate the MAD based on improvement of subjective complaints. The actual mechanism of titration will be individually trained with each patient.
2. Titration during drug-induced sleep endoscopy (DISE) - DISE-assisted titration:

   The DISE will be performed by an ear-nose-throat (ENT)surgeon experienced in DISE in order to visualize the dose-dependent effect of the mandibular protrusion on the upper airway collapsibility. The DISE is performed in a semi-dark and silent operating theatre with the patient lying in supine position. The different collapsible levels of the upper airway that can be investigated during DISE are the palate (velopharynx), the oropharynx, the tongue base, the hypopharynx and the epiglottis. The degree of collapse at each level is reported as none, partial or complete. The pattern of the pharyngeal collapse during the obstructive events are classified as concentric, anteroposterior and/or laterolateral. Upon connection of the RCMP to a dedicated laptop, calibration of the actual versus the software-guided protrusion is verified using the RCMP ruler and proprietary developed software, to rule out day-to-day variation caused by environmental factors such as room temperature or humidity. This procedure ensures the mandibular displacement to be read out correctly from the ruler present at the upper tray fitted over the tooth arcs. After the calibration, the RCMP-trays are fitted in edge-to-edge position to avoid excessive muscle tension. A flexible fibreoptic nasendoscope will be introduced by the ENT surgeon in the awake patient to evaluate the awake upper airway state. Thereafter, sedation will be induced by intravenous administration of midazolam (bolus injection of 1.0 to 2.0 mg) and propofol using a target-controlled infusion system (2.0 to 3.0 μg/mL). The transition to unconsciousness similar to stage 2 sleep is aimed at and examined by assuring absence of patients' eyelash reflex after stimulation by means of a gentle brush. Findings are noted using a uniform upper airway scoring system evaluating level of snoring, presence of apneas and degree of oxygen saturation, degree and configuration of obstruction(s) and the level of upper airway collapse. When target sedation is reached, examined by assuring absence of patients' eyelash reflex after stimulation by means of a gentle brush, the RCMP will be remotely protruded in increments of 2 mm in response to the visualized upper airway collapse at the different collapsible levels until a stable upper airway together with absence of desaturations and snoring is reached. If a stable upper airway in absence of snoring is noted, oxygen desaturation and apneas are evaluated, and the mandible will be remotely retruded for 1 mm. If the upper airway remains stable, further so-called 'reversed titration' will continue. This approach will be repeated until the effective target protrusive position can be determined, defined as the minimal mandibular threshold position corresponding to a stable upper airway in the absence of snoring, oxygen desaturation and apneas. When a stable upper airway is reached, the titration procedure will be continued in 0.5 mm steps, to be as precise as possible. After every protrusive or retrusive movement the RCMP protrusion will be checked on the RCMP ruler versus the protrusion measured by the software, assuring correct positioning of the mandible during the upper airway evaluation.
3. Titration during polysomnography (PSG):

At the start of the PSG, the participant's dental trays are attached to the mandibular positioner of the RCMP device, and the positioner is calibrated to the PSG system using the device software. The titration procedure that will be used in this study is previously described. Once asleep, the patient's mandible will be protruded remotely in 0.5 mm steps in response to evidence of apneas and/or hypopneas. If an EEG arousal occurs, no further advancement will be attempted until stable sleep resumes. Stepwise mandibular protrusion will continue until respiratory events are reduced to normal in all sleep stages, and in both supine and lateral position, or until maximal protrusion is reached. Afterwards, an independent researcher will score the PSG together with body position and mandibular position signals and will predict success or failure with MAD therapy based on the predetermined interpretative rules. The patient needs to have rapid eye movement (REM) sleep for ≥ 5 minutes in the supine position or in the lateral position, if REM in supine position was not observed. All REM cycles will be evaluated to identify a minimum 5 minutes' interval where ≤ 1 respiratory event occurred. If this is the case, the PSG will be scored as predicted MAD success for that protrusive position. If not, the PSG will be judged to predict therapeutic failure. The predicted effective target protrusive position is the minimum protrusive position that is associated with ≤ 1 respiratory event per 5-minutes REM interval. If the PSG is scored as predicted success, the predicted effective target protrusive position is provided to the dentist to start MAD therapy in that position. If the PSG is scored as predicted failure, an alternative position equal to 75% of maximal protrusion is provided.

A polygraphic evaluation of the MAD efficacy will be planned after each titration procedure. Furthermore, the patients will be asked to fill out questionnaires regarding snoring, daytime sleepiness (Epworth Sleepiness Scale, ESS), fatigue (Checklist Individual Strength, CIS20R) and side effects of the MAD treatment.

A wash-out period of one week is inserted between the polygraphic evaluation of the protrusive position obtained during a titration procedure and the start of the next titration procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe obstructive sleep apnea (OSA) (obstructive AHI (oAHI) ≥ 15/h)
* BMI < 30 kg/m²
* Age > 18 year
* PSG < 2 years old with stable body weight (+/- 5 kg), no ENT surgery since most recent PSG and stable clinical condition
* Normal clinical and radiological (incl. OPG), periodontal en temporomandibular joint examination
* Subject is capable of giving informed consent
* No documented abuses (alcohol, drugs, …)

Exclusion Criteria:

* Edentulous patients
* Insufficient teeth to support the mandibular advancement device
* Active periodontal problems including tooth mobility
* Active temporomandibular joint dysfunction
* Limited maximum protrusive capacity (<6 mm)
* Limited vertical opening (<25 mm)
* Enlarged palatine tonsils (Grade IV tonsils)
* Degenerative neuromuscular disorders
* Pregnancy or willing to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-04-07 (Actual)

PRIMARY OUTCOMES:
The amount of protrusion (mm) | After the patient underwent the three titration procedures, so approximately 4 months after start of the study
  The protrusive position that was predicted as the effective target protrusive position during each titration method (subjective titration, RCMP titration PSG and RCMP titration DISE) will be assessed and compared between the different titration methods.

SECONDARY OUTCOMES:
The apnea/hypopnea index (AHI) derived from the polysomnographic evaluation. | After the patient underwent the three titration procedures, so approximately 4 months after start of the study
  The efficacy of the MAD therapy will be assessed as a measure of treatment outcome by comparingthe baseline AHI with the AHI under MAD therapy.

OTHER OUTCOMES:
Visual analogue scale for snoring | After the patient underwent the three titration procedures, so approximately 4 months after start of the study
  A standard 10-point visual analogue scale (VAS) ranging from 0 to 10 with 0 equaling no snoring and 10 causing the bed partner to leave the room or sleep separately was used to evaluate the subjective status of snoring, as assessed by the bed partner. Heavy snoring was defined as a VAS snoring index of at least 7. A decrease of at least 3 points on VAS for snoring during treatment with MAD compared to baseline represents a decrease of one level of snoring severity and was therefore considered satisfactory. To be considered as an important'important' reduction, snoring had to be reduced to a snoring index that was no longer evaluated as bothersome, i.e. to a snoring index of ≤ 3.
Epworth sleepiness scale | After the patient underwent the three titration procedures, so approximately 4 months after start of the study
  Hypersomnolence was assessed using the Epworth Sleepiness Scale (ESS), an 8-item questionnaire which takes about three minutes to fill out. It reflects the chance of each person's general level of sleepiness during eight situations of daily life. The subject selects the most appropriate integer score ranging from 0 (would never doze) to 3 (high chance of dozing) for each of the 8 questions. The results are then summed up, with 0 being the minimal and 24 the maximum total ESS score. The higher the ESS score, the higher that person's average sleep propensity in daily life. In general, ESS scores need to be interpreted as follows: 0-5=Lower Normal Daytime Sleepiness, 6-10 = Higher Normal Daytime Sleepiness, 11-12 = Mild Excessive Daytime Sleepiness, 13-15 = Moderate Excessive Daytime Sleepiness, 16-24 =Severe Excessive Daytime Sleepiness.
Checklist Individual Strenght | After the patient underwent the three titration procedures, so approximately 4 months after start of the study
  Fatigue severity was assessed using the Checklist Individual Strength (CIS20R), a 20-item questionnaire that takes around five to ten minutes to fill out. Each question has a statement to be scored on a 7-point Likert scale ranging between 'yes, this is true' to 'no, this is not true'. The total score is calculated as the sum of the responses to the different statements. The maximum CIS20R score is 140, with a score of 76/140 or higher indicating that the patient is at risk for prolonged absence at work. The scale is subdivided in four dimensions of fatigue being fatigue severity (8 items, max. score 56), concentration problems (5 items, max. score 35), reduced motivation (4 items, max. score 28) and activity (3 items, max. score 21).

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Vanderveken, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University of Antwerp, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dieltjens M, Braem MJ, Op de Beeck S, Vroegop AVMT, Kazemeini E, Van de Perck E, Beyers J, Kastoer C, Wouters K, Willemen M, Verbraecken JA, Vanderveken OM. Remotely controlled mandibular positioning of oral appliance therapy during polysomnography and drug-induced sleep endoscopy compared with conventional subjective titration in patients with obstructive sleep apnea: protocol for a randomized crossover trial. Trials. 2019 Oct 29;20(1):615. doi: 10.1186/s13063-019-3698-4. PMID 31665059